CLINICAL TRIAL: NCT06945328
Title: Study of Patients With Drug-induced Non-variceal Upper Gastrointestinal Bleeding
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Abdelfattah Ahmed, Principal investigator, Assiut University
Other Study IDs: Gastrointestinal Bleeding
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Upper Gastrointestinal Bleeding (UGIB)
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Upper endoscopy — All patients will do gastroscopy (upper endoscopy) within the first 24 hour of admission and specific elements of bleeding

SUMMARY:
* To study the association between non-variceal UGIB and the use of NSAIDs, VKAs, DOACs and antiplatelet therapy.
* To compare the severity of bleeding related to specified drugs.
* To determine risk factors associated with non-variceal UGIB.

DETAILED DESCRIPTION:
Upper gastrointestinal bleeding (UGIB) carries a high mortality, especially in elderly patients having co-morbidities, and the incidence of non-variceal and variceal bleeding is reported to be 3.5% and 15%, respectively.

Atrial fibrillation, deep vein thrombosis, pulmonary embolism, and other conditions require anticoagulation, non-steroidal anti-inflammatory drugs (NSAIDs) and antiplatelet therapy putting the patients at high risk of hemorrhage.

The latest American Heart Association (AHA) report on cardiovascular diseases suggests a doubling of the prevalence of atrial fibrillation by 2030 compared to 2010. The need to institute anticoagulation for this condition, both as primary and secondary prevention, will automatically increase the number of UGIB cases. An improvement in this regard has occurred with the advent of direct oral anticoagulants (DOACs) which have been shown to be non-inferior to vitamin K antagonists (VKAs).

In the event of UGIB, the Rockall score is a valid prediction score, repeatedly confirmed to assess the risk of patients with non-variceal bleeding. The management of UGIB is commonly adapted according to this score. Identifying high-risk patients who may benefit from longer hospitalization is crucial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years and above) presented with signs and symptoms of UGIB (hematemesis and/or melena)

Exclusion Criteria:

* Variceal bleeding
* Age below 18 years
* Pregnant women
* Consent refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 18 years and above) presented either to the emergency or the outpatient department with signs and symptoms of UGIB (hematemesis and/or melena) who are on the specified medications (NSAIDs, VKAs, DOACs and antiplatelet therapy).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Association between non-variceal UGIB and the use of different drugs | through study completion, an average of 1 year
  observation the association between the incedience of Non-variceal upper Gastrointestinal Bleeding and the use of NSAIDs, VKAs, DOACs and antiplatelet therapy

SECONDARY OUTCOMES:
The severity of Non-variceal bleeding related to specified drugs. | through study completion, an average of 1 year
  To compare the severity of Non-variceal bleeding related to specified drugs, according to Rockall Score
Risk factors associated with non-variceal upper gastrointestinal bleeding | through study completion, an average of 1 year
  We will determine risk factors associated with With non-varicreal gastrointestinal bleeding, such as demographic data, smoking , co-morbidities ، dose and duration of specified drugs, and presence of h pylori infection.

REFERENCES:
- [Background] Kim BJ, Park MK, Kim SJ, Kim ER, Min BH, Son HJ, Rhee PL, Kim JJ, Rhee JC, Lee JH. Comparison of scoring systems for the prediction of outcomes in patients with nonvariceal upper gastrointestinal bleeding: a prospective study. Dig Dis Sci. 2009 Nov;54(11):2523-9. doi: 10.1007/s10620-008-0654-7. Epub 2008 Dec 23. PMID 19104934
- [Background] Rockall TA, Logan RF, Devlin HB, Northfield TC. Influencing the practice and outcome in acute upper gastrointestinal haemorrhage. Steering Committee of the National Audit of Acute Upper Gastrointestinal Haemorrhage. Gut. 1997 Nov;41(5):606-11. doi: 10.1136/gut.41.5.606. PMID 9414965
- [Background] Sjogren V, Bystrom B, Renlund H, Svensson PJ, Oldgren J, Norrving B, Sjalander A. Non-vitamin K oral anticoagulants are non-inferior for stroke prevention but cause fewer major bleedings than well-managed warfarin: A retrospective register study. PLoS One. 2017 Jul 10;12(7):e0181000. doi: 10.1371/journal.pone.0181000. eCollection 2017. PMID 28700711
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Background] Piran S, Schulman S. Treatment of bleeding complications in patients on anticoagulant therapy. Blood. 2019 Jan 31;133(5):425-435. doi: 10.1182/blood-2018-06-820746. Epub 2018 Dec 17. PMID 30559261
- [Background] Piccini JP, Hellkamp AS, Lokhnygina Y, Patel MR, Harrell FE, Singer DE, Becker RC, Breithardt G, Halperin JL, Hankey GJ, Berkowitz SD, Nessel CC, Mahaffey KW, Fox KA, Califf RM; ROCKET AF Investigators. Relationship between time in therapeutic range and comparative treatment effect of rivaroxaban and warfarin: results from the ROCKET AF trial. J Am Heart Assoc. 2014 Apr 22;3(2):e000521. doi: 10.1161/JAHA.113.000521. PMID 24755148
- [Background] Ullrich H, Gori T. Antiplatelet therapies in patients with an indication for anticoagulation. Clin Hemorheol Microcirc. 2016;64(3):273-278. doi: 10.3233/CH-168104. PMID 28128753
- [Background] Steffel J. Stroke Prevention with Non-Vitamin K Oral Anticoagulants: For Most, but Not for All! Cardiology. 2019;143(3-4):121-123. doi: 10.1159/000501586. Epub 2019 Jul 26. No abstract available. PMID 31352454
- [Background] Hearnshaw SA, Logan RF, Lowe D, Travis SP, Murphy MF, Palmer KR. Acute upper gastrointestinal bleeding in the UK: patient characteristics, diagnoses and outcomes in the 2007 UK audit. Gut. 2011 Oct;60(10):1327-35. doi: 10.1136/gut.2010.228437. Epub 2011 Apr 13. PMID 21490373
- [Background] Targownik LE, Nabalamba A. Trends in management and outcomes of acute nonvariceal upper gastrointestinal bleeding: 1993-2003. Clin Gastroenterol Hepatol. 2006 Dec;4(12):1459-1466. doi: 10.1016/j.cgh.2006.08.018. Epub 2006 Nov 13. PMID 17101296